CLINICAL TRIAL: NCT02420808
Title: An Epidemiological Cohort Study of Acute Coronary Syndromes in The Greek Population. The PHAETHON Study
Acronym: PHAETHON
Status: Completed | Type: Observational
Sponsor: Hellenic Cardiovascular Research Society (Other)
Responsible Party: Sponsor
Other Study IDs: PHAETHON
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease
Keywords: CAD; STEMI; non STEMI; Unstable angina; Greece
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A nationwide registry of patients with acute coronary disease to evaluate epidemiological patient characteristics, medical management, implementation of invasive strategy, patient outcome and impact on quality of life in Greece.

DETAILED DESCRIPTION:
A nationwide registry of patients with acute coronary disease to evaluate epidemiological patient characteristics, medical management, implementation of invasive strategy, patient outcome and impact on quality of life in Greece.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* > 25 years
* Admission in hospital within 24 hours from beginning of symptoms of transfer from antother hospital within 24 hours from beginning of symptoms.
* Acute Coronary Syndrom

Exclusion Criteria:

-

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ACS
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of patients with Acute Coronary Syndromes. | 6 months
  Assessment of the epidemiological characteristics of patients who were hospitalized with a diagnosis of ACS. Evaluation of the therapeutic strategy and its outcome.

SECONDARY OUTCOMES:
Estimation of the percentage of patients. | Baseline
  Estimation of the percentage of patients who were hospitalized with STEMI, NSTEMI and unstable angina.
Description of the methods of patients' evacuation. | Baseline
  Description of the methods of patients' evacuation from the scene of the incident to the receiving hospital where was processed the treatment for ACS.
Estimation of the interval until the arrival in the hospital. | Baseline
  Estimation of the duration from the onset of pain until the arrival in the receiving hospital at various locations.
Evaluation of the blood test analysis during hospitalization. | Baseline
  Evaluation of hematological, biochemical parameters and myocardial necrosis markers during hospitalization.
Description of the administered medication. | Baseline - 6 months
  Description of the pharmaceutical treatment administered during hospitalization and monitoring period.
Evaluation of the male patients with erectile dysfunction. | Baseline - 6 months
  Estimation of the percentage of the male patients with erectile dysfuction based to a predesigned questionnaire and investigation of the possible association with the treatment's outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Chalkida, Chalcis, Greece